CLINICAL TRIAL: NCT03121794
Title: Ultrasonographic Identification of the Proximal Humerus Landmarks for Intra-Osseous Vascular Access Across Different Body Habitus
Brief Title: Ultrasonographic Identification of the Proximal Humerus Landmarks
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, SergioB17, Principal Investigator, The Cleveland Clinic
Other Study IDs: 16-1642
Record Dates: First submitted 2017-03-23; First posted 2017-04-20 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-08

CONDITIONS: Proximal Humerus Interosseous Venous Access; Anatomic Landmark; Ultrasonography
Keywords: ultrasonography; Intraosseous Vascular access; humerus; anatomic landmark

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Low BMI: Ultrasonographic identification of proximal humerus landmarks for patients with BMI 18.5 - 25 kg/m2
  Interventions: Procedure: Ultrasonographic exam; Device: ultrasound machine
- Moderate BMI: Ultrasonographic identification of proximal humerus landmarks for patients with BMI 30-35 kg/m2 will receive ultrasound exam.
  Interventions: Procedure: Ultrasonographic exam; Device: ultrasound machine
- High BMI: Ultrasonographic identification of proximal humerus landmarks for patients with BMI > 40 kg/m2 will receive ultrasound exam.
  Interventions: Procedure: Ultrasonographic exam; Device: ultrasound machine

INTERVENTIONS:
Procedure: Ultrasonographic exam — The study team will perform an ultrasonographic exam of the proximal humerus to identify six anatomical landmarks
Device: ultrasound machine — Regular ultrasound machine used at Cleveland Clinic

SUMMARY:
Evaluate whether discrete landmarks of the proximal humerus can be identified using ultrasound in patients with various body habitus and BMI.

DETAILED DESCRIPTION:
There are three main forms of vascular access: peripheral intravenous (PIV), Central venous (CV) and intraosseous (IO). Of the different types of vascular access PIV and CV access have drawbacks when used during resuscitation, because they can be difficult to obtain when patients are volume depleted as in cases of trauma. Attempting CV access has numerous risks with complications occurring in up to 33% of attempts. These include failed placement (22%), arterial puncture (5%), catheter malposition (4%), pneumothorax (1%) and asystolic cardiac arrest (<1%). Attempting to obtain CV access may also disrupt chest compressions in cases of cardiac arrest. Intraosseous access has been used in scenarios where PIV and CV access is difficult or impossible to obtain. Pharmacokinetic studies and standard practice support the bioequivalence of intraosseous and intravenous administration of common medications. Intravascular depletion does not hinder attempts at IO access, and as the insertion sites are peripheral to the heart, insertion can be done avoiding interruptions in chest compressions. Obtaining proximal humerus interosseous (PHIO) access may also be faster than obtaining both PIV and CV access with a relatively low complication rate. In one survey, complications of IO included difficulty in identifying correct anatomical site (3%), extravasation (3.7%), displacement after insertion (8.5%), and very rarely late complications including compartment syndrome (0.6%), osteomyelitis (0.4%) and skin infection (0.3%).

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older undergoing general, cardiac, thoracic or vascular surgery.
* BMI >= 18.5 kg/m^2

Exclusion Criteria:

* Limited mobility/ range of motion of arms
* Prior surgical intervention on shoulder or humerus
* History of arm dislocation with internal rotation
* History of arm fracture
* BMI in ranges: 25.1 - 29.9, 35.1 - 39.9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected after chart review of current patients undergoing general, cardiac, thoracic, or vascular surgery. Patients will be approached in the preoperative clinic or during their hospitalization (preoperatively or postoperatively). Informed consent will be obtained prior to performing the study.
  Participants will be separated into 3 cohorts based on BMI. The number of participants in each cohort is as follows: 10 patients with BMI 18.5 - 25 kg/m2; 10 patients with BMI 30-35 kg/m2, 10 patients with BMI > 40 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Number of proximal humerus landmarks successfully identified by ultrasound exam | Through completion of ultrasonographic exam, an average of 30 minutes.
  Two investigators will perform an ultrasonographic exam on each patient, with one investigator examining each side of the body. Each investigator will aim to identify 6 anatomical landmarks:
  1. The humeral shaft,
  2. The surgical neck of the humerus,
  3. The lesser tubercle,
  4. The greater tubercle,
  5. The intertubercular sulcus
  6. The target site in the greater tubercle for needle insertion. Each side will receive a score ranging from 0 to 6 corresponding to the number of landmarks correctly identified.

SECONDARY OUTCOMES:
Time used to identify all 6 anatomical landmarks using ultrasound in seconds. | Through completion of ultrasonographic exam, an average of 30 minutes.
  Evaluate the time used to identify all 6 anatomical landmarks using ultrasound.
Depth of each landmark from the skin in centimeters. | Through completion of ultrasonographic exam, an average of 30 minutes.
  Depth of each landmark from the skin in centimeters based on ultrasound measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT03121794/Prot_SAP_000.pdf